CLINICAL TRIAL: NCT00916513
Title: Quality of Life and Treatment Satisfaction of People With Type 2 Diabetes: A European Survey
Acronym: PANORAMA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Other Study IDs: NIS-CEU-DUM-2008/2
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes
Keywords: Diabetes; Treatment Satisfaction; Quality of Life; HbA1c levels and goals; Healthcare resources consumption
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients ³ 40 years old, with T2DM diagnosed and followed up in the participating site at least 1 year prior to entry in the study, treated with diet, OADs and/or insulin for at least the past three months

SUMMARY:
The present European survey seeks to assess quality of life and satisfaction with treatment in people with T2DM and to appreciate disease and treatment variables including hypoglycaemia and level of glycaemic control. It will also provide relevant information on other important aspects such as the level of correlation of objective measures such as HbA1c with health status, QoL and satisfaction with current treatment. Overall 5000 randomly selected patients will be invited to participate from a representative sample of clinical practices during a pre-specified period. The study will entail a single patient visit. Patients who agree to the study and give their informed consent will complete questionnaires which, combined with retrospective notes review & an HbA1c test, will allow patient, disease and treatment variables to be collected. An HbA1c test is a finger prick test to measure glycosylated haemoglobin in the blood indicating the level of blood glucose over the last 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* With T2DM, diagnosed at least 1 year prior to entry in the study
* Currently treated with diet, OAD(s) and/or insulin with no change in the type of OAD(s) or insulin in the previous three months

Exclusion Criteria:

* Type 1 diabetes and/or history of diabetic ketoacidosis
* Secondary diabetes (including disease of the exocrine pancreas, endocrinopathies or drug-induced)
* Treatment with systemic glucocorticoids other than replacement therapy. Inhaled, local injected and topical use of glucocorticoids is allowed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be recruited in Primary Care Centres mainly, but hospitals will be allowed in some countries
Sampling Method: Probability Sample
Enrollment: 5926 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Diabetes-related QoL and treatment satisfaction questionnaires: DTSQ, ADDQoL, HFSws and EQ5D | Cross-sectional and retrospective

SECONDARY OUTCOMES:
Disease-related variables: Years with diabetes, use of SMBG and frequency of monitoring, Hypoglycaemic episodes, Past Medical History, Macro and micro-vascular complications | Retrospective (previous 24 months)
Health-economic variables: Use of healthcare resources Days off work (for either hypoglycaemias, acute or chronic complications) | Retrospective (previous 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles Porta, Study Director — Medical Department.AstraZeneca Spain
Locations (302):
- France (176):
  - Research Site, Antibes
  - Research Site, Athies
  - Research Site, Audruicq
  - Research Site, Auxerre
  - Research Site, Baigneux-les-Juifs
  - Research Site, Baume-les-Dames
  - Research Site, Beaumont-sur-Lèze
  - Research Site, Beaurepaire
  - Research Site, Beauvais
  - Research Site, Bettacourt La Ferree
  - Research Site, Bezons
  - Research Site, Bérat
  - Research Site, Béziers
  - Research Site, Blois
  - Research Site, Boulogne-sur-Gesse
  - Research Site, Bresles
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Bruère-Allichamps
  - Research Site, Bulles
  - Research Site, Burry
  - Research Site, Cany-Barville
  - Research Site, Capdenac-Gare
  - Research Site, Cappelle-Brouck
  - Research Site, Carquefou
  - Research Site, Carresse-Cassaber
  - Research Site, Carros
  - Research Site, Celles-sur-Plaine
  - Research Site, Champagnole
  - Research Site, Champigny-sur-Marne
  - Research Site, Chanmpdeniers Saint Denis
  - Research Site, Chartrettes
  - Research Site, Chauvigny
  - Research Site, Châbons
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Clairac
  - Research Site, Clichy
  - Research Site, Comps
  - Research Site, Concarneu
  - Research Site, Courbevoie
  - Research Site, Courpière
  - Research Site, Coutances
  - Research Site, Coutouvre
  - Research Site, Dambach-la-Ville
  - Research Site, Dieulouard
  - Research Site, Digoin
  - Research Site, Donges
  - Research Site, Douchy-les-Mines
  - Research Site, Drap
  - Research Site, Escaudain
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Faverges
  - Research Site, Fenouillet
  - Research Site, Firmi
  - Research Site, Francoville La Garenne
  - Research Site, Fruges
  - Research Site, Gelles
  - Research Site, Gondrecourt-le-Château
  - Research Site, Guitalens-L'Albarède
  - Research Site, Hanvec
  - Research Site, Houilles
  - Research Site, Hyères
  - Research Site, Ivry-sur-Seine
  - Research Site, Jussey
  - Research Site, L'Haÿ-les-Roses
  - Research Site, La Courneuve
  - Research Site, La Crau
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Mulatière
  - Research Site, La Tranche-sur-Mer
  - Research Site, Lamagistère
  - Research Site, Lanouaille
  - Research Site, Laroquebrou
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Le Cannet
  - Research Site, Le Grand-Lemps
  - Research Site, Le Havre
  - Research Site, Le Monastier-sur-Gazeille
  - Research Site, Le Nouvion-en-Thiérache
  - Research Site, Le Pertre
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Pontet
  - Research Site, Les Mées
  - Research Site, Leyme
  - Research Site, Lézignan-Corbières
  - Research Site, Locmiquélic
  - Research Site, Luneray
  - Research Site, Lyon
  - Research Site, Magland
  - Research Site, Maintenon
  - Research Site, Mantes-la-Ville
  - Research Site, Marcq-en-Barœul
  - Research Site, Marles-les-Mines
  - Research Site, Marseille
  - Research Site, Mauléon-Licharre
  - Research Site, Mayet
  - Research Site, Meximieux
  - Research Site, Mezzavia
  - Research Site, Miramas
  - Research Site, Monce En Berlin
  - Research Site, Montélimar
  - Research Site, Montfort-en-Chalosse
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montreuil
  - Research Site, Monts-sur-Guesnes
  - Research Site, Mussidan
  - Research Site, Narbonne
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Nice
  - Research Site, Niederschaeffolsheim
  - Research Site, Noisy-le-Sec
  - Research Site, Nordausques
  - Research Site, Nouâtre
  - Research Site, Oberhausbergen
  - Research Site, Orchies
  - Research Site, Orliénas
  - Research Site, Ormes
  - Research Site, Pantin
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pauillac
  - Research Site, Pernes-les-Fontaines
  - Research Site, Pibrac
  - Research Site, Pierrepont-sur-Avre
  - Research Site, Pitgam
  - Research Site, Plancoët
  - Research Site, Pléneuf-Val-André
  - Research Site, Plouvorn
  - Research Site, Pornic
  - Research Site, Port-La Nouvelle
  - Research Site, Pradines
  - Research Site, Puilley Les Vignes
  - Research Site, Puttelange-aux-Lacs
  - Research Site, Quessoy
  - Research Site, Quiberon
  - Research Site, Quimper
  - Research Site, Rambervillers
  - Research Site, Renazé
  - Research Site, Richemont
  - Research Site, Robion
  - Research Site, Romainville
  - Research Site, Rombas
  - Research Site, Romorantin-Lanthenay
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-Aubin-des-Châteaux
  - Research Site, Saint-Bonnet-le-Château
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Saëns
  - Research Site, Saint-Thuriau
  - Research Site, Saint-Yorre
  - Research Site, Salles
  - Research Site, Salomé
  - Research Site, Sassenage
  - Research Site, Sault-lès-Rethel
  - Research Site, Soissons
  - Research Site, Soisy-sur-École
  - Research Site, Soyaux
  - Research Site, Ste Menehould
  - Research Site, Strasbourg
  - Research Site, Thann
  - Research Site, Thuré
  - Research Site, Toufflers
  - Research Site, Toulon
  - Research Site, Tourcoing
  - Research Site, Troyes
  - Research Site, Uzès
  - Research Site, Vailly-sur-Aisne
  - Research Site, Valenton
  - Research Site, Valras-Plage
  - Research Site, Vaugneray
  - Research Site, Villefagnan
  - Research Site, Villejuif
  - Research Site, Villeurbanne
  - Research Site, Vitry-le-François
- Germany (48):
  - Research Site, Aachen
  - Research Site, Alsdorf
  - Research Site, Ampfing
  - Research Site, Aschersleben
  - Research Site, Augsburg
  - Research Site, Bad Freienwalde
  - Research Site, Bad Staffelstein
  - Research Site, Berlin
  - Research Site, Biberbach
  - Research Site, Bonn
  - Research Site, Coburg
  - Research Site, Duisburg
  - Research Site, Edenkoben
  - Research Site, Erfurt
  - Research Site, Eschweiler
  - Research Site, Essen
  - Research Site, Frechen
  - Research Site, Fuchsstadt
  - Research Site, Fulda
  - Research Site, G�ntersleben
  - Research Site, Hamburg
  - Research Site, Heinsberg
  - Research Site, Holzkirchen
  - Research Site, Homburg
  - Research Site, Iserlohn
  - Research Site, Kaisersesch
  - Research Site, Kalkar
  - Research Site, Kehl
  - Research Site, Kirchheim
  - Research Site, Klingenberg
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Marpingen
  - Research Site, Moers
  - Research Site, München
  - Research Site, Nuremberg
  - Research Site, Oberursel
  - Research Site, Pretzfeld
  - Research Site, Reit im Winkl
  - Research Site, Rimbach
  - Research Site, Sand
  - Research Site, Schwaig
  - Research Site, Sinntal
  - Research Site, Sonthofen
  - Research Site, Westerkappeln
  - Research Site, Wiesbaden
  - Research Site, Zweibrücken
  - Research Site, Zwenkau
- Research Site, Athens, Greece
- Ireland (2):
  - Research Site, Belfast
  - Research Site, Co. Anrtim
- Italy (4):
  - Research Site, Andria, Bari
  - Research Site, Latina
  - Research Site, Rome
  - Research Site, Viterbo
- Netherlands (36):
  - Research Site, Beilen, Drenthe
  - Research Site, Coevorden, Drenthe
  - Research Site, Zwartemeer, Drenthe
  - Research Site, Almere Stad, Flevoland
  - Research Site, Lichtenvoorde, Gelderland
  - Research Site, Nijmegen, Gelderland
  - Research Site, Maastricht, Limburg
  - Research Site, Vlodorp, Limburg
  - Research Site, 's-Hertogenbosch, Noord-Braband
  - Research Site, Beek en Donk, Noord-Braband
  - Research Site, Etten-Leur, Noord-Braband
  - Research Site, Lieshout, Noord-Braband
  - Research Site, Schijndel, Noord-Braband
  - Research Site, Soerendonk, Noord-Braband
  - Research Site, Edam, North Holland
  - Research Site, Hoogwoud, North Holland
  - Research Site, Huizen, North Holland
  - Research Site, Volendam, North Holland
  - Research Site, Ermelo, Overijssel
  - Research Site, Heeten, Overijssel
  - Research Site, Hengelo, Overijssel
  - Research Site, Nijverdal, Overijssel
  - Research Site, Tubbergen, Overijssel
  - Research Site, Drachten, Provincie Friesland
  - Research Site, Onstwedde, Provincie Groningen
  - Research Site, Bennebroek, South Holland
  - Research Site, Dordrecht, South Holland
  - Research Site, Lisse, South Holland
  - Research Site, Rijswijk, South Holland
  - Research Site, Roelofarendsveen, South Holland
  - Research Site, Rotterdam, South Holland
  - Research Site, Spijkernisse, South Holland
  - Research Site, The Hague, South Holland
  - Research Site, Woerden, South Holland
  - Research Site, Amersfoort, Utrecht
  - Research Site, Poortvliet, Zeeland
- Spain (11):
  - Research Site, Cadiz, Andalusia
  - Research Site, Santander, Cantabria
  - Research Site, Burgos, Castille and León
  - Research Site, Manresa, Catalonia
  - Research Site, Barcelona, Catalu�a
  - Research Site, Pontevedra, Galicia
  - Research Site, Gran Canaria, Las Palmas de Gran Canaria
  - Research Site, Coslada, Madrid
  - Research Site, Fuenlabrada, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Elche, Valencia
- United Kingdom (24):
  - Research Site, Bath
  - Research Site, Bedford
  - Research Site, Birmingham
  - Research Site, Blackburn
  - Research Site, Blackpool
  - Research Site, Bristol
  - Research Site, Bury St Edmunds
  - Research Site, Cambridge
  - Research Site, Canterbury
  - Research Site, Cardiff
  - Research Site, Cornwall
  - Research Site, Coventry
  - Research Site, Darlington
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, Penzance
  - Research Site, Plymouth
  - Research Site, Reading
  - Research Site, Salisbury
  - Research Site, Sheffield
  - Research Site, St Albans

REFERENCES:
- [Derived] Bradley C, Eschwege E, de Pablos-Velasco P, Parhofer KG, Simon D, Vandenberghe H, Gonder-Frederick L. Predictors of Quality of Life and Other Patient-Reported Outcomes in the PANORAMA Multinational Study of People With Type 2 Diabetes. Diabetes Care. 2018 Feb;41(2):267-276. doi: 10.2337/dc16-2655. Epub 2017 Nov 28. PMID 29183910
- [Derived] Simon D, de Pablos-Velasco P, Parhofer KG, Gonder-Frederick L, Duprat Lomon I, Vandenberghe H, Eschwege E, Bradley C. Hypoglycaemic episodes in patients with type 2 diabetes--risk factors and associations with patient-reported outcomes: The PANORAMA Study. Diabetes Metab. 2015 Dec;41(6):470-9. doi: 10.1016/j.diabet.2015.08.007. Epub 2015 Oct 9. PMID 26455870
- [Derived] de Pablos-Velasco P, Parhofer KG, Bradley C, Eschwege E, Gonder-Frederick L, Maheux P, Wood I, Simon D. Current level of glycaemic control and its associated factors in patients with type 2 diabetes across Europe: data from the PANORAMA study. Clin Endocrinol (Oxf). 2014 Jan;80(1):47-56. doi: 10.1111/cen.12119. Epub 2013 May 6. PMID 23194193
- [Derived] Bradley C, de Pablos-Velasco P, Parhofer KG, Eschwege E, Gonder-Frederick L, Simon D. PANORAMA: a European study to evaluate quality of life and treatment satisfaction in patients with type-2 diabetes mellitus--study design. Prim Care Diabetes. 2011 Dec;5(4):231-9. doi: 10.1016/j.pcd.2011.04.004. Epub 2011 Jul 14. PMID 21752743